CLINICAL TRIAL: NCT01496963
Title: Observational Multicenter Study Lasting 12 Months to Determine the Prevalence of Pulmonary Hypertension (PAH) in Patients With Thalassemia Major and Intermedia and Verify the Suitability of Common Diagnostic Criteria in This Population
Brief Title: Prevalence of Pulmonary Hypertension (PAH) in Patients With Thalassemia
Acronym: PAH2010
Status: Completed | Type: Observational
Sponsor: Ente Ospedaliero Ospedali Galliera (Other)
Responsible Party: Principal Investigator, Dr. Gian Luca Forni, Principal Investigator and Chief of Centre for Microcythemia an Congenital Anemias - Hematology, Ente Ospedaliero Ospedali Galliera
Other Study IDs: PAH2010
Record Dates: First submitted 2011-12-14; First posted 2011-12-22 (Estimated); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Thalassemia Major; Thalassemia Intermedia; Pulmonary Arterial Hypertension
Keywords: Thalassemia; Pulmonary Arterial Hypertension
MeSH Terms: conditions — beta-Thalassemia; Pulmonary Arterial Hypertension; Thalassemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- group a): Patients with pulmonary artery pressure (PAP) assessed (by echocardiogram) <36 mmHg or a tricuspid regurgitant jet velocity (TG) <3 m / sec and data on PAP and mean left ventricular ejection fraction (LVEF) > 50%
  Interventions: Other: Physician standard-of-care according to ESC/ERS Guidelines
- group b): Patients with:
  PAP estimated (by echocardiography)> 40 mmHg or TG> 3.2 m / sec and LVEF> 50% As indicated by the Guidelines, patients b) with increased PAP (TG> 3.2 m / sec or> 40 mm Hg) will be further studied using RHC and vasoreactivity testing. Angio CAT, 6MWT and BNP.
  Interventions: Other: Physician standard-of-care according to ESC/ERS Guidelines
- group c): patients with PAP estimated (by echocardiography) in the range of values > 3 m / sec (TG) and <3.2 m / sec or> 36 mm Hg and <40 mmHg and LVEF> 50%
  Interventions: Other: Physician standard-of-care according to ESC/ERS Guidelines

INTERVENTIONS:
Other: Physician standard-of-care according to ESC/ERS Guidelines — Physician standard-of-care

SUMMARY:
This is a multicenter observational case-control analysis lasting 12 months aimed at determining the prevalence of pulmonary hypertension (PAH) in patients with Thalassemia Major and Intermedia. The patients will be followed, treated and examined according to the best standard clinical practice dictated by the Italian Society for the study of Hemoglobinopathies (SITE), Thalassemia International Federation (TIF)and the Task Force for Diagnosis and Treatment of Pulmonary Hypertension of European Society of Cardiology (ESC); European Respiratory Society (ERS); International Society of Heart and Lung Transplantation (ISHLT) guidelines.

DETAILED DESCRIPTION:
The most recent International Classification of pulmonary arterial hypertension (PHA) include Hemoglobinopathies in Class I. At present there is no determination of the prevalence of this disease in a large population of thalassemic patients followed in a uniform way. The diagnostic criteria used for the normal population may not be suitable for a population such as thalassemia patients who present features like chronic anemia, iron overload, liver disease, endocrine disorders, etc.

The criteria used to define the disease (PHA) will be those ones dictated by the above mentioned guidelines.

Primary Objective of the study is the determination of the prevalence and severity of PHA in thalassemia syndromes, recently introduced in Class I of the Classification of PHA.

Secondary objectives are:

Critical evaluation of current diagnostic criteria derived from those applied to the general population, taking into account the peculiarities of the observed disease in the thalassemic population.

Evaluation of sensitivity and specificity of echocardiogram versus right cardiac catheterization (RHC).

Evaluation of the correlation between:

echocardiography and RHC; resistance and heart rate determined both by RHC and echocardiography; Determination of the patients resulted vasoreactive during RHC. Validation of sensitivity and specificity (sens/spec) of 6 minutes walking test (6MWT) and brain natriuretic peptide (BNP) in Thalassemia Major (TM) and Intermediate (TI) with reference to specific pulmonary hypertensive disease

In order to achieve the objectives of the study observed patients will be divided into group according to the following the criteria:

group a)

* Pulmonary artery pressure (PAP) assessed (by echocardiogram) < 36 mmHg or a tricuspid regurgitant jet velocity (TG) < 3 m/sec and data on PAP and mean left ventricular ejection fraction (LVEF) > 50% group b)
* PAP estimated (by echocardiography)> 40 mmHg or TG > 3.2 m / sec and LVEF> 50%
* As indicated by the Guidelines, patients b) with increased PAP (TG > 3.2 m / sec or > 40 mm Hg) will be further studied using RHC and vasoreactivity testing. Angio CAT, 6MWT and BNP.

group c) - PAP estimated (by echocardiography) in the range of values > 3 m/sec (TG) and < 3.2 m / sec or > 36 mm Hg and <40 mmHg and LVEF > 50% Each case included both in group b) and c) will be paired with two controls included in the group a) to make the groups more comparable.

The group a) will serve as control group to compare the diagnostic methods evaluated as per protocol.

In order to divide the patients into the three groups specified above first it will be evaluated: PAP, LVEF% and TG assessed by echocardiographic examination performed in the six months prior to the beginning of the study (thalassemic patients have to perform echocardiography once a year to monitor cardiac function according to the guidelines)

Patients belonging to groups a), b) and c) will perform the following assessments:

- Clinical cardiac evaluation according to the New York Heart Association (NYHA) (functional class I to IV)

As per the International Guidelines, patients belonging to groups b) and c) have clinical indications to undergo Two-dimensional echocardiography-Doppler Duplex Scanner (PW) and color flow (CW) to determine the following parameters:

* End-systolic volume and left ventricular end diastolic, indexed according to body surface
* Percentage change of right ventricular areas (area diastolic/systolic area expressed as a percentage%)
* Tricuspid lateral annulus excursion Longitudinal (TAPS)
* Eccentricity Index (EI)
* TG
* Pulmonary resistance.

Moreover, patients belonging to group b), according to the International Guidelines have clinical indication to undergo RHC, diagnostic evaluation to rule out the presence of associated diseases and to measure:

* Pulmonary pressures
* Mean atrial pressure
* Pulmonary resistance
* Cardiac rate
* Vasoreactivity test

To compare the data derived from the RHC and the echocardiography the following echocardiographic parameters will be further evaluated:

Right atrial pressure; Cardiac output; Pulmonary wedge pressure

ELIGIBILITY:
Inclusion Criteria:

* Patients with Thalassemia Major Patients or Intermediate referring to Centres using Web-Thal medical record (a clinical data sheet used for congenital anemias. Info: www.thalassemia.it)

Exclusion Criteria:

* Patients who are considered potentially unreliable and/or not cooperative

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Thalassemia Major and Intermedia studied by echocardiography in the six months prior to the beginning of the study
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2012-01; Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Determination of the prevalence | 12 months
  Determination of the prevalence, defined as the total number of cases in the population, divided by the number of individuals in the population.

SECONDARY OUTCOMES:
Critical evaluation of current diagnostic criteria | 12 months
  Critical evaluation of current diagnostic criteria taking into account the peculiarities of the observed of PHA in thalassemic patients.

CONTACTS AND LOCATIONS:
Locations (8):
- Italy (8):
  - SCDU Microcitemie-Pediatria A.O. Universitaria S.Luigi Gonzaga di Orbassano, Orbassano, Turin
  - Divisione di Ematologia Ospedale Perrino, Brindisi
  - Clinica pediatrica Ospedale Microcitemico, Cagliari
  - DH Microcitemia dell'adulto Ospedale Microcitemico, Cagliari
  - Centro della Microcitemia e delle Anemie Congenite -Ematologia e Cardiologia E.O. Ospedali Galliera, Genoa
  - Centro Anemie Congenite Università di Milano IRCCS Ospedale Maggiore Policlinico, Milan
  - Dipartimento di pediatria "F.Fede" A.O. Universitaria FedericoII di Napoli, Napoli
  - U.O.C- Cardiologia Ospedale San Francesco, Nuoro

REFERENCES:
- [Background] Task Force for Diagnosis and Treatment of Pulmonary Hypertension of European Society of Cardiology (ESC); European Respiratory Society (ERS); International Society of Heart and Lung Transplantation (ISHLT); Galie N, Hoeper MM, Humbert M, Torbicki A, Vachiery JL, Barbera JA, Beghetti M, Corris P, Gaine S, Gibbs JS, Gomez-Sanchez MA, Jondeau G, Klepetko W, Opitz C, Peacock A, Rubin L, Zellweger M, Simonneau G. Guidelines for the diagnosis and treatment of pulmonary hypertension. Eur Respir J. 2009 Dec;34(6):1219-63. doi: 10.1183/09031936.00139009. Epub 2009 Sep 12. No abstract available. PMID 19749199
- [Derived] Derchi G, Galanello R, Bina P, Cappellini MD, Piga A, Lai ME, Quarta A, Casu G, Perrotta S, Pinto V, Musallam KM, Forni GL; Webthal Pulmonary Arterial Hypertension Group*. Prevalence and risk factors for pulmonary arterial hypertension in a large group of beta-thalassemia patients using right heart catheterization: a Webthal study. Circulation. 2014 Jan 21;129(3):338-45. doi: 10.1161/CIRCULATIONAHA.113.002124. Epub 2013 Sep 30. PMID 24081970